CLINICAL TRIAL: NCT03287141
Title: Comparison of CPAP and Bi-level Effects on Exercise Tolerance and Cardiorespiratory Responses in Individuals With Chronic Heart Failure.
Brief Title: CPAP Versus Bi-level in Chronic Heart Failure
Acronym: CHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patri-cia Angelica de Miranda Silva Nogueira (Other)
Responsible Party: Sponsor-Investigator, Patri-cia Angelica de Miranda Silva Nogueira, PhD, Universidade Federal do Rio Grande do Norte
Organization: Universidade Federal do Rio Grande do Norte (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1a2b3c4d
Record Dates: First submitted 2017-09-12; First posted 2017-09-19 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Heart Failure
Keywords: noninvasive ventilation; continuous positive airway pressure; intermittent positive-pressure breathing; exercise test; physical endurance; physical fitness
MeSH Terms: conditions — Heart Failure | interventions — Walk Test; Noninvasive Ventilation; Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First intervention (Sham Comparator): The subjects did a shuttle walk test without any previous intervention.
  Interventions: Diagnostic Test: Shuttle walk test
- Second intervention (Experimental): Subjects underwent 30 minutes of noninvasive ventilation (CPAP) and then re-performed the shuttle walk test.
  Interventions: Device: Noninvasive ventilation (CPAP)
- Third intervention (Experimental): Subjects underwent 30 minutes of noninvasive ventilation (Bi-pap) and then re-performed the shuttle walk test.
  Interventions: Device: Noninvasive ventilation (Bi-pap)

INTERVENTIONS:
Diagnostic Test: Shuttle walk test — A shuttle walk test was performed without any previous intervention.
  Arms: First intervention
Device: Noninvasive ventilation (Bi-pap) — After 30 minutes of the mentioned intervention, the subject performed a shuttle walk test.
  Arms: Third intervention
Device: Noninvasive ventilation (CPAP) — After 30 minutes of the mentioned intervention, the subject performed a shuttle walk test.
  Arms: Second intervention

SUMMARY:
Introduction: Dyspnea and fatigue are the main clinical symptoms of heart failure and primarily responsible for exercise intolerance found in this syndrome. Now, It is known that the use of NIV in CPAP mode applied before exercise increases exercise tolerance in people with heart failure; however, it's not yet known if the bi-level mode is able to generate similar or even better results, due to pressure increase of the ventilatory support in this modality. Moreover, it is possible that there is influence between the pressure levels set in the NIV and the magnitude of its effect on the exercise in this population Objective: 1) test for differences between the acute effects of NIV on exercise tolerance in patients with HF, when applied CPAP or bi-level mode; and 2) check for discrepancies in the acute effects of Bi-level mode on the physical performance of these individuals, when applied at different pressure levels. Methodology: This is a controlled, randomized, double-blind and cross-over clinical trial, to be composed of 45 volunteers of both genders, aged between 30 and 80 years, with chronic heart failure, functional class II and III (New York Heart Association) in clinical stability. The experiment will be carried out on four different days, with a 48-hour interval between them, in which NIV will be used in the following modes: Bi-level with minimum parameters (EPAP = 6 cmH2O and IPAP = 12 cmH2O), Bi-level with maximum parameters EPAP = 8 cmH2O and IPAP = 14 cmH2O) and CPAP (6 cmH2O). Thus, all the volunteers will participate in the four TGC. During the tests, distance walking, perceived levels of fatigue and dyspnea, affective response, as well as other physiological variables will be analyzed. Statistical analysis, the ANOVA test for repeated measurements will be used, followed by the Bonferroni post-test, considering p-value less than or equal to 0.05 as statistically significant. Expected Results: This work is expected to improve the therapeutic management of HF patients, assisting in the implementation and improvement of methods to improve dyspnea and muscle fatigue, thus increasing tolerance to exercise.

DETAILED DESCRIPTION:
This study is a randomized controlled trial, double-blind and cross-over, to be composed of 45 volunteers of both genders, aged between 30 and 80 years, with CHF will be selected from a specialized outpatient clinic with medical consent. Patients should have symptoms of compensated CHF; presenting functional capacity II and III (New York Heart Association), with left ventricular ejection fraction <50%; not participating in cardiac rehabilitation programs; and clinical stability in the last three months, with no history of angina or coexistence of obstructive pulmonary disease (Tiffeneau-Pinelli index> 70% in spirometry). In addition, they should not present any osteoarticular or neurological disease would prevents them from performing the proposed tests, as well as having a score higher than 22 in the Leganés cognitive test (20). In the case of NIV or exercise intolerance, as well as in case of non-attendance to the experiments on the scheduled days, subjects will be excluded from the study.

The sample will be the result of a non-probabilistic sampling process, calculated based on the magnitude of the effect of the main variable (distance traveled) after the use of NIV therapy, obtained in a pilot study. In addition, this protocol was aproved by the institution's Ethics Committee on Human Research (CAAE: 49324415.0.000.5537).

Experimental procedure The experimental protocol will occur in three visits, one per day, with a minimum interval of 48 hours between them. On the first visit, the volunteers will undergo a screening that consists of clinical evaluation (assessment sheet) and cognitive (Leganéscognitive test), as well as evaluation of lung function (spirometry) and QoL (Minnesota Living with Heart Failure Questionnaire). Next, the Shuttlel Walking Test (SWT) control (T-Co) will be performed, without previous use of NIV, in order to determine the distance traveled and other physiological variables in the absence of interventions. Finally, during the initial visit, a preliminary NIV session will be held to adjust the interface and adapt the volunteer to the therapy.

At each subsequent visit, volunteers will perform a SWT immediately after 30 minutes of NIV, one day in Bi-level mode and one in CPAP mode, following a randomized sequence. Thus, all volunteers will perform one SWT after CPAP (T-CP) and one SWT after Bi-level (T-Bi). In the experiment, the CPAP pressure will be maintained at 6 cmH2O, while at the Bi-level an expiratory pressure (EPAP) of 6 cmH2O and an inspiratory pressure (IPAP) of 12 cmH2O will be defined.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient and have a compensated HF, without hospitalizations in the last three months;
2. Present functional class II and III (New York Heart Association);
3. Present left ventricular ejection fraction (LVEF) ≤ 50%;
4. Have not suffered myocardial infarction in the last three months;
5. No previous diagnosis of chronic obstructive pulmonary disease (FEV1 / FVC ratio> 70% in spirometry);
6. Do not be a smoker;
7. Not being pregnant;
8. Does not present any clinical disease or restriction of osteomioarticular or neurological origin that prevents / limits the carrying out of the proposed tests;
9. Integral cognitive functions, which were evaluated by the cognitive test of Leganés - PCL

Exclusion Criteria:

1. Unstable angina or significant arrhythmias;
2. Acute atrial fibrillation or total atrioventricular block;
3. Systemic blood pressure (AP) at uncontrolled rest (≥ 180/110 mmHg or ≤80 / 40mmHg);
4. Resting heart rate (HR) ≤ 40 bpm or ≥ 120 bpm;
5. Need for dialysis;
6. Use of bronchodilator;
7. Respiratory rate (RF) at rest ≥ 35 rpm;
8. Frequent vomiting;
9. Intolerance to NIV;
10. infection or fever.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10-19; Primary Completion 2015-11-23 (Actual); Study Completion 2016-03-23 (Actual)

PRIMARY OUTCOMES:
Physical exercise tolerance | Immediately after the test
  The distance covered in the shuttle walk test

SECONDARY OUTCOMES:
Perception of effort | before and immediately after the test
  The muscular fatigue of the legs
Perception of dyspnea | before and immediately after the test
  The discomfort in the breath
Respiratory rate | before and immediately after the test
  The number of times an individual breathed in a minute.
Peripheral oxygen saturation | before and immediately after the test
  Noninvasive measurement of peripheral oxygen saturation by re-evaluating oxygenation rate.
Heart rate | before and immediately after the test
  Heart rate reflecting heart beats for one minute.
Blood pressure | before and immediately after the test
  Variable blood pressure analysis performed noninvasively.

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia Nogueira, PhD, Principal Investigator — college professor

IPD SHARING:
Plan to Share IPD: Undecided